CLINICAL TRIAL: NCT06058585
Title: The Chronic Kidney Disease Adaptive Platform Trial Investigating Various Agents for Therapeutic Effect
Acronym: CAPTIVATE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P01351; U1111-1324-3113 (Other: World Health Organisation, Universal Trial Number (UTN))
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic kidney disease; Mineralocorticoid Receptor Antagonist; Finerenone
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — finerenone

STUDY DESIGN:
Intervention Model Description: Adaptive platform trial evaluating multiple interventions in multiple domains of therapeutic care. Additional interventions and participants will be added as the trial grows.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The default position within CAPTIVATE is that treatment allocations determined by randomisation will be provided on a blinded basis. Blinding, however, may not always be feasible particularly for behavioural or device-related interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Finerenone (Experimental): Finerenone 10mg or 20mg tablets
  Interventions: Drug: Finerenone
- Placebo Finerenone (Placebo Comparator): Finerenone matched placebo tablets
  Interventions: Drug: Placebo Finerenone

INTERVENTIONS:
Drug: Finerenone — Finerenone 10mg or 20mg tablets, oral, once daily
  Other Names: BAY94-8862
  Arms: Finerenone
Drug: Placebo Finerenone — Finerenone matched placebo tablets, oral, once daily
  Arms: Placebo Finerenone

SUMMARY:
CAPTIVATE is an international, multi-centre, Phase III, adaptive, platform, randomised controlled trial in people with chronic kidney disease (CKD).

CAPTIVATE aims to find the best treatment, or combination of treatments, that slow the progression of CKD so that fewer people develop kidney failure.

CAPTIVATE provides a research platform that allows many treatment-related questions to be answered within a common trial set-up.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) affects over 800 million people globally and is projected to be the 5th most common cause of death by 2040. CKD progresses to kidney failure, increases the risk of early death, heart disease, and leads to a poorer quality of life.

Current treatments do not entirely remove the risk of kidney failure in people with CKD. To improve the outcomes of people with CKD, it is crucial to find the best treatment or combination of treatments that can slow CKD progression. CAPTIVATE aims to address this need.

CAPTIVATE has been designed to test multiple treatments within a common research platform. This design is more efficient and will lead to a shorter time for patients to receive effective treatments. The trial is 'eternal', which means that participants will continue to be recruited for many years until the trial is finally wound up. It is also 'adaptive', providing the flexibility to add new treatments, or remove those that are not working.

Participants can participate in more than one treatment at the same time or at different times. Participants receive each study treatment for 2 years. For each treatment, participants are followed up at study visits that occur at approximately one month, 3 months, 6 months, 12 months, 18 months and 2 years after starting treatment. A final study visit occurs one month after the end of the 2-year treatment phase. Information collected at study visits include blood and urine test results, safety assessments and treatment adherence. Information about the overall health status of each participant is collected every 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Known chronic kidney disease from any cause (eGFR ≥25 mL/min/1.73m2)
3. Currently receiving standard of care treatment according to treating physician
4. Eligible for randomisation in at least one recruiting domain-specific appendix
5. Participant and treating physician are willing and able to perform trial procedures

Exclusion Criteria:

1. Planned to commence kidney replacement therapy or kidney transplant surgery in next 6 months
2. Life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
eGFR slope | From randomisation to week 108
  eGFR slope calculated using eGFR values from randomisation to week 108

SECONDARY OUTCOMES:
Change in albuminuria | From randomisation to week 24
  Change in albuminuria as measured by uACR (or uPCR if uACR unavailable) between randomisation and 24 weeks, measured as a continuous variable
Composite of 40% eGFR decline or kidney failure | From randomisation to week 108
  Composite outcome of proportion of participants experiencing a 40% eGFR decline between randomisation and 108 weeks, and proportion of participants developing kidney failure (defined as eGFR <15 mL/min/1.73m2 or chronic kidney replacement therapy start) at 108 weeks
All-cause mortality at 108 weeks | 108 weeks
  Incidence of death from any cause
Number of cardiovascular events | 108 weeks
  Number of cardiovascular events (cardiovascular death, hospitalised heart failure, myocardial infarction, stroke)
Safety and tolerability of treatment | 108 weeks
  Incidence and rates of adverse events, and time from commencement of study treatment until interruption of treatment due to toxicity.
Change in quality of life | From randomisation to week 108
  Change in quality of life measured using the Quality of Life Impact Survey for Kidney Disease (QDIS-CKD) at 6-monthly intervals from randomisation to week 108

CONTACTS AND LOCATIONS:
Overall Officials: Sradha Kotwal, Study Chair — The George Institute; Hiddo Lambers Heerspink, Study Chair — The George Institute
Locations (32):
- Australia (13):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Nepean Blue Mountains Local Health District, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast Hospital and Health Service, Birtinya, Queensland
  - Townsville University Hospital, Douglas, Queensland
  - West Moreton Hospital & Health Service, Ipswich, Queensland
  - Gold Coast Hospital and Health Service, Southport, Queensland
  - Royal Adelaide, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Austin Health, Heidelberg, Victoria
  - South Metropolitan Health Service, Fiona Stanley Hospital, Murdoch, Western Australia
- India (13):
  - Gitam Institute of Medical Sciences and Research, Visakhapatnam, Andhra Pradesh
  - Patna Medical College and Hospital, Patna, Bihar
  - Father Muller Medical College Hospital, Mangaluru, Karnataka
  - Dr Moopen's Medical College, Meppādi, Kerala
  - CARE-CHL Hospital, Indore, Madhya Pradesh
  - Medway Hospital, Chennai, Tamil Nadu
  - Yashoda Hospital Hitec City, Hyderabad, Telangana
  - Apollo Hospitals, Hyderabad, Telangana
  - Charak Hospital and Research Centre, Lucknow, Uttar Pradesh
  - Shri Guru Ram Rai Medical College and Shri Mahant Indiresh Hospital, Dehradun, Uttarakhand
  - Fortis Hospital, Kolkata, West Bengal
  - North Bengal Medical College & Hospital, Siliguri, West Bengal
  - Max Superspeciality Hospital, Dehradun, Dehradun
- New Zealand (6):
  - Health New Zealand, Te Whatu Ora Te Matau a Maui, Hawke's Bay Hospital, Hastings, Hawkes Bay
  - Health New Zealand, Te Whatu Ora Waitemata, North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland
  - Aotearoa Clinical Trials Trust, Middlemore Hospital, Auckland
  - 201 Great King Street, Central Dunedin, Dunedin 9016, New Zealand, Dunedin
  - Private Bag 9742 Maunu Road, Horahora, Whangārei 0148, New Zealand, Whangarei

IPD SHARING:
Plan to Share IPD: Yes
Trial data will be made available as a resource for future unspecified research, subject to any prior contractual obligations. Researchers wishing to gain access to the study resources will be required to submit an application for review by the Platform Oversight Committee, including a detailed project description, a list of data requested, and evidence of ethical approval. De-identified data extracts will be made available to approved proposals, and will not include data obtained from data linkage with local registries.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: TBC
Access Criteria: Assessments of data requests will be based on sound science, benefit-risk balancing and research team expertise.

REFERENCES:
- [Derived] Kotwal SS, Perkovic V, Jardine MJ, Kim D, Shah NA, Lin E, Coggan S, Billot L, Vart P, Wheeler DC, de Boer IH, Zhang H, Hou FF, Sugawara Y, Marion J, Lewis RJ, Berry LR, McGlothlin A, Jha V, De Nicola L, Gorriz JL, Heerspink HJL; GKPTN and CAPTIVATE Investigators. The Global Kidney Patient Trials Network and the CAPTIVATE Platform Clinical Trial Design: A Trial Protocol. JAMA Netw Open. 2024 Dec 2;7(12):e2449998. doi: 10.1001/jamanetworkopen.2024.49998. PMID 39661388
- [Derived] Heerspink HJL, Kretzler M. Clinical Trials for Kidney Disease in the Era of Personalized Medicine. J Am Soc Nephrol. 2024 Aug 1;35(8):1123-1126. doi: 10.1681/ASN.0000000000000412. Epub 2024 May 9. No abstract available. PMID 39248631